CLINICAL TRIAL: NCT02638727
Title: Assessment of Short-term Effect of L-Citrulline on Endothelial Function and Vasodilation in Known CAD Patients:A Randomized Crossover Clinical Trial
Brief Title: Assessment of Short-term Effect of L-Citrulline on Endothelial Function and Vasodilation in Known CAD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Ali Akbarzadeh, sistant proffesor of shahid beheshti university of medical sciences, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CVRC101
Record Dates: First submitted 2015-11-08; First posted 2015-12-23 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Vascular Disease
Keywords: vascular disease; endothelial function; L-Citrulline
MeSH Terms: conditions — Vascular Diseases | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Drug Arm (Active Comparator): This group treat with L-Citrulline (3 grams per day)
  Interventions: Drug: L-Citrulline
- Placebo Arm (Placebo Comparator): this group treat with placebi every day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: L-Citrulline — This group treat with L-Citrulline (3 grams per day)
  Arms: Drug Arm
Drug: placebo — This group treat with placebo dayley
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to determine the efficacy of oral L-Citrulline on endothelial function and vasodilation in patients with coronary artery disease(CAD) by evaluating the brachial artery diameter in the antecubital area by ultrasonography.

DETAILED DESCRIPTION:
Before prescribing the drug or placebo, the patients were evaluated via the ultrasound machine equipped. The brachial artery diameter in the antecubital area was measured by the ultrasound and was recorded. Then blood pressure cuff was attached on the arm and dilated 50mmhg above the systolic pressure and for 5 minutes remained the same level to induce ischemia at distal tissues until the occurrence of compensatory vasodilatation. Then the brachial artery diameter (as an estimation of FMD) was measured and recorded. After 4 minutes of administration of 2 puffs of nitroglycerin spray, the brachial artery diameter (as an estimation of NMD) was measured.

After 15 days treatment with the L-Citrulline or the placebo, the patients underwent the ultrasonography again and the above assessments were done.

Improvement of FMD to NMD ratio (before L-Citrulline prescription) to FMD to NMD ratio (after L-Citrulline prescription) is determined as "improvement of flow mediated dilation to nitroglycerin dependent vasodilation" evaluate.

ELIGIBILITY:
Inclusion Criteria:

* history of documented CAD; flow mediated dilation to nitroglycerin dependent vasodilation (FMD/NMD)ratio less than 1

Exclusion Criteria:

* no documented CAD; flow mediated dilation to nitroglycerin dependent vasodilation (FMD/NMD)ratio equal /more than 1

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
improvement of flow mediated dilation to nitroglycerin dependent vasodilation | 15 days
  improvement of FMD to NMD ratio (before L-Citrulline prescription) to FMD to NMD ratio (after L-Citrulline prescription)

CONTACTS AND LOCATIONS:
Overall Officials: Morteza Safi, MD, Study Director — Cardiovascular Research Center
Locations (1):
- Shahid Modaress Hospital , Tehran, Iran, Tehran, Iran